CLINICAL TRIAL: NCT05448651
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Multiple Ascending-Dose Study to Assess the Safety, Tolerability, Immunogenicity, Pharmacokinetics and Pharmacodynamics of UPB-101 in Subjects With Asthma
Brief Title: Safety and Biologic Impact (Pharmacodynamics) of Repeated Injections and Increasing Amounts of UPB-101 in Asthmatics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Upstream Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UPB-CP-01
Record Dates: First submitted 2022-06-29; First posted 2022-07-07 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active substance 1 (Experimental): UPB-101 Cohort 1
  Interventions: Drug: UPB-101; Drug: Placebo
- Active substance 2 (Experimental): UPB-101 Cohort 2
  Interventions: Drug: UPB-101; Drug: Placebo
- Active substance 3 (Experimental): UPB-101 Cohort 3
  Interventions: Drug: UPB-101; Drug: Placebo
- Active Substance 4 (Experimental): UPB-101 Cohort 4
  Interventions: Drug: UPB-101; Drug: Placebo

INTERVENTIONS:
Drug: UPB-101 — Subcutaneous injection
  Other Names: Formerly ASP7266
Drug: Placebo — Subcutaneous injection
  Other Names: 0.9% saline solution

SUMMARY:
The goals of this clinical study were to assess the safety, tolerability, blood levels, and disease impact of UPB-101 when given to adults with mild asthma. Eligible participant were consecutively assigned to 1 of 3 to 5 planned treatment groups. Each treatment group consisted of 8 individuals, six of whom will received active drug (UPB-101) and 2 who received placebo. Neither the study doctors nor the participants knew which participants were assigned to active study drug and which were assigned to placebo. The study was performed at 4 experienced research sites in the United Kingdom.

DETAILED DESCRIPTION:
This was a two-part phase 1b, multi-center randomized, double-blind (Investigator and Subject blinded; Sponsor unblinded), placebo-controlled, multiple ascending-dose study to assess the safety, tolerability, immunogenicity, pharmacokinetics (PK), and pharmacodynamics (PD) of UPB-101 administered subcutaneously (SC) to adult subjects with asthma.

The study consists of Part A and Part B. Part A included 3 cohorts with pre-set dosing regimens. Part B (optional) included up to 2 additional cohorts whose doses and dosing intervals decided based upon the safety, PK, and PD results from Part A (i.e., an adaptive design), as applicable. The regimens selected for Part B did not exceed the exposures (i.e., doses and/or dosing intervals) included in Part A. Eight subjects were randomized per cohort (6 active, 2 placebo). Thus, a total of 32 subjects were enrolled in the study with 24 subjects in Part A and 8 in Part B.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 to 60, and has physician-diagnosed asthma
2. Body mass index (BMI) between 18 and 35 kg/m2
3. Blood eosinophil cell count ≥200 (OR ≥150 combined with fractional exhaled nitric oxide [a measure of lung airway inflammation] >25) at one screening visit and ≥150 at the other screening
4. Agrees to follow the required contraceptive techniques
5. Female or male participant agrees not to donate eggs or sperm, respectively, for a period of 120 days after the last dose of the study drug
6. Able to perform spirometry (breathing tests)
7. Asthma and non-biologic asthma medication have been stable for the past 2 months

Exclusion Criteria:

1. Employee, consultant, and/or immediate family member of any person involved in the conduct of the study
2. Previous exposure to the study drug or known allergy/sensitivity to any of its ingredients
3. Pregnant or breastfeeding female
4. Unable to fast and avoid strenuous exercise for 9 hours prior to each site visit
5. Serious allergic reaction to any injected drug
6. Significantly abnormal clinical laboratory test results or a significant medical condition
7. Recently donated blood (including blood products) or experienced significant loss of blood
8. Has pacemaker or a significantly abnormal electrocardiogram
9. An active or a serious infection in the past 8 weeks
10. Poorly-controlled diabetes or abnormal kidney function
11. Tests positive to illicit drugs or nicotine and cannot limit alcohol consumption
12. Tests positive for human immunodeficiency virus antibodies (HIV), hepatitis B, hepatitis C antibodies, or tuberculosis
13. Received any vaccine within the past month
14. Received any immunosuppressant therapies in the past
15. Received an antibody or therapeutic biologic product in the last 6 months
16. Received steroids (other than inhaled) in the past 2 months
17. Participated recently in a clinical study
18. Current tobacco smokers or has smoked within the last year
19. Tested positive for COVID-19 in the past month

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sumathi Sivapalasingam, MD, Study Director — Upstream Bio
Locations (4):
- United Kingdom (4):
  - Hammersmith Medicines Research, London
  - Queen Anne Street Medical Centre, London
  - Richmond Pharmacology, London
  - Medicines Evaluation Unit, Manchester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 4 sites in the United Kingdom (UK).
Groups:
- Active Substance 1: UPB-101 Cohort 1 (100 mg)
- Active Substance 2: UPB-101 Cohort 2 (200 mg)
- Active Substance 3: UPB-101 Cohort 3 (300 mg)
- Active Substance 4: UPB-101 Cohort 4 (25 mg)
Period: Overall Study
Arm/Group | Active Substance 1 | Active Substance 2 | Active Substance 3 | Active Substance 4 | Placebo
Started | 6 | 6 | 6 | 6 | 8
Completed | 6 | 6 | 6 | 6 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Substance 1 | Active Substance 2 | Active Substance 3 | Active Substance 4 | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (10.31) | 37.7 (8.82) | 32.7 (9.54) | 48.0 (5.25) | 37.0 (11.41) | 38.1 (10.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 2 | 2 | 3 | 16
  Male | 1 | 2 | 4 | 4 | 5 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 5 | 6 | 6 | 6 | 7 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 3 | 0 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1 | 2
  White | 4 | 4 | 2 | 6 | 7 | 23
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 6 | 6 | 6 | 8 | 32
BMI at Screening (kg/m2) [Mean (Standard Deviation); unit: kg/m^2] | 26.57 (3.025) | 25.18 (2.074) | 25.22 (2.848) | 27.65 (2.518) | 25.56 (3.110) | 26.01 (2.784)

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-emergent Adverse Events and Serious Adverse Events
Description: Overall Summary of Treatment-emergent Adverse Events (TEAEs) and Adverse Events (AEs) up to Week 24 (Safety Population)
Time Frame: Baseline through 24 weeks
Measure: Number; unit: adverse events
Arm/Group | Active Substance 1 | Active Substance 2 | Active Substance 3 | Active Substance 4 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
adverse events
  any TEAEs | 19 | 17 | 12 | 9 | 25
  SAEs | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Incidence of Anti-drug Antibodies
Description: Blood samples were analyzed for the presence of ADAs using validated assays. Low titer ADA responses were detected toward the end of the concentration vs time profile. There was no evident effect of ADAs on drug exposure and no immune-related adverse events
Time Frame: Baseline through Week 32
Population: Subjects who received any kind of study intervention, and had at least one blood sample measured for ADAs.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Substance 1 | Active Substance 2 | Active Substance 3 | Active Substance 4 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
Participants | 4 | 5 | 1 | 2 | 0

3. Secondary Outcome: Maximum Observed Concentration of UPB-101
Description: Blood samples were collected and analyzed using a validated assay to determine the Cmax (ug/mL) of UPB-101. The pharmacokinetic (PK) parameters were estimated using non-compartmental analysis.
Time Frame: First Dose = Day 1. Last Dose = Baseline through 32 weeks.
Population: The PK Population included all subjects who received at least 1 complete dose of active study drug (UPB-101) and for whom at least 1 PK parameter was estimated.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Active Substance 1 | Active Substance 2 | Active Substance 3 | Active Substance 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
ug/mL
  Cmax after first dose | 8.82 (2.25) | 21.8 (3.78) | 32.4 (6.23) | 1.85 (0.602)
  Cmax after last dose: number analyzed (Participants) | 4 | 4 | 6 | 0
  Cmax after last dose | 16.3 (5.03) | 41.8 (5.69) | 33.8 (8.39) |

4. Secondary Outcome: Time to Maximum Observed Concentration of UPB-101
Description: Blood samples were collected and analyzed using a validated assay to determine the Tmax (days) of UPB-101. The pharmacokinetic (PK) parameters were estimated using non-compartmental analysis.
Time Frame: Baseline through 32 weeks
Population: as for outcome 3
Measure: Median (Full Range); unit: days
Arm/Group | Active Substance 1 | Active Substance 2 | Active Substance 3 | Active Substance 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
days
  Tmax after first dose | 6.98 [2.92 to 14.0] | 5.95 [2.77 to 13.9] | 6.93 [5.93 to 6.98] | 9.94 [2.90 to 20.9]
  Tmax after last dose: number analyzed (Participants) | 4 | 4 | 6 | 0
  Tmax after last dose | 5.00 [2.99 to 7.04] | 3.94 [2.90 to 6.91] | 4.98 [2.91 to 13.9] |

5. Secondary Outcome: Area Under the Concentration-time Curve Under One Dosing Interval of UPB-101
Description: Blood samples were collected and analyzed using a validated assay to determine the AUClast (d.ug/mL) of UPB-101. The pharmacokinetic (PK) parameters were estimated using non-compartmental analysis.
Time Frame: Baseline through 32 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Active Substance 1 | Active Substance 2 | Active Substance 3 | Active Substance 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
day*μg/mL
  AUClast after the first dose | 187 (40.8) | 449 (101) | 1220 (236) | 73.4 (26.6)
  AUClast after the last dose: number analyzed (Participants) | 4 | 4 | 6 | 0
  AUClast after the last dose | 613 (115) | 1740 (496) | 1420 (453) |

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Treatment-emergent Adverse Events Reported by at Least 5% of Participants Overall up to Week 24 (Safety Population)
Arm/Group | Active Substance 1 | Active Substance 2 | Active Substance 3 | Active Substance 4 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 5/6 | 6/6 | 5/6 | 3/6 | 6/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Substance 1 (N=6) | Active Substance 2 (N=6) | Active Substance 3 (N=6) | Active Substance 4 (N=6) | Placebo (N=8)
Rhinitis (Infections and infestations) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 3 (3)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Asthma exercise induced (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (5) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menopausal symptoms (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/51/NCT05448651/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-17): https://cdn.clinicaltrials.gov/large-docs/51/NCT05448651/SAP_001.pdf